CLINICAL TRIAL: NCT04118621
Title: Role of Chest Ultrasound in Detection of Post-operative Pulmonary Complications After Cardiothoracic Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ali zein elabdein abd elaleim, principle investigator, Assiut University
Other Study IDs: chest ultrasound after CTS
Record Dates: First submitted 2019-09-26; First posted 2019-10-08 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: IHD; Valve Heart Disease; Surgery--Complications
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: chest ultrasound — detection of postoperative pulmonary complications after cardiothoracic surgery

SUMMARY:
* assess feasibility of detecting pulmonary complications postoperative using chest ultrasound compared to chest x-ray
* measure time lag between using ultrasound and using chest x-ray to detect pulmonary complications postoperative

DETAILED DESCRIPTION:
It is well known that cardiothoracic surgery causes different types of pulmonary complications like residual pleural effusion and pneumothorax therefore it is common that surgeons make a thoracic drainage by introducing intercostal tubes for evacuation of air and fluid from the pleural space. Complications extend to involve the parenchymal pulmonary tissue causing consolidation or involve the interstitial tissue .all these complications affect the postoperative recovery.

As a classical technique a daily chest X-ray is performed from first day of surgical intervention to hospital discharge to assess the amount of residual pleural effusion so drainage removal can be done or not and also assess other pulmonary complications.

However, chest X-rays are costly, exposing patients and health care workers to ionizing radiation requiring patient movement with chest drains, difficult positioning of the patient to get good films, and time consuming.

On the other hand, using chest ultrasound is a good alternative for chest X-ray because it is a bedside, easier, more sensitive and accurate in detection of pulmonary complications.

Its main advantages represented in avoiding the danger of ionizing radiations, easier device portability, low cost and a rapid learning curve.

So it is easy and less time consuming to correlate between ultrasound findings and clinical data and assist in invasive procedures.

Hypothesis that detecting pulmonary complications postoperative using chest ultrasound is easier, more sensitive and accurate compared to chest X-ray.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cardiothoracic surgery at Assiut University Hospital include CABG, Valve replacement, minimal invasive cardiac surgeries, thoracic surgeries as open thoracotomy and VATS surgeries and others.
* Age >18yrs: 80yrs.

Exclusion Criteria:

* Patients <18yr and >80yrs.
* patient refused to be enrolled in research
* patient with subcutaneous emphysema

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiothoracic surgery at Assiut University Hospital who meet the listed inclusion, include CABG, Valve replacement, minimal invasive cardiac surgeries, thoracic surgeries as open thoracotomy and VATS surgeries and others
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
detecting pulmonary complications postoperative using chest ultrasound compared to chest x-ray | 1 week
  assess feasibility of detecting pulmonary complications postoperative using chest ultrasound compared to chest x-ray as chest ultrasound is easier, more sensitive and accurate

REFERENCES:
- [Background] Amorosa JK, Bramwit MP, Mohammed TL, Reddy GP, Brown K, Dyer DS, Ginsburg ME, Heitkamp DE, Jeudy J, Kirsch J, MacMahon H, Ravenel JG, Saleh AG, Shah RD. ACR appropriateness criteria routine chest radiographs in intensive care unit patients. J Am Coll Radiol. 2013 Mar;10(3):170-4. doi: 10.1016/j.jacr.2012.11.013. PMID 23571057
- [Background] Graham RJ, Meziane MA, Rice TW, Agasthian T, Christie N, Gaebelein K, Obuchowski NA. Postoperative portable chest radiographs: optimum use in thoracic surgery. J Thorac Cardiovasc Surg. 1998 Jan;115(1):45-50; discussion 50-2. doi: 10.1016/s0022-5223(98)70441-6. PMID 9451044
- [Background] Leschber G, May CJ, Simbrey-Chryselius N. [Do thoracic surgery patients always need a postoperative chest X-ray?]. Zentralbl Chir. 2014 Sep;139 Suppl 1:S43-9. doi: 10.1055/s-0034-1383034. Epub 2014 Sep 29. German. PMID 25264723
- [Background] Chung MJ, Goo JM, Im JG, Cho JM, Cho SB, Kim SJ. Value of high-resolution ultrasound in detecting a pneumothorax. Eur Radiol. 2005 May;15(5):930-5. doi: 10.1007/s00330-004-2518-7. Epub 2004 Dec 18. PMID 15609058
- [Background] Soni NJ, Franco R, Velez MI, Schnobrich D, Dancel R, Restrepo MI, Mayo PH. Ultrasound in the diagnosis and management of pleural effusions. J Hosp Med. 2015 Dec;10(12):811-6. doi: 10.1002/jhm.2434. Epub 2015 Jul 28. PMID 26218493
- [Background] Vezzani A, Manca T, Brusasco C, Santori G, Valentino M, Nicolini F, Molardi A, Gherli T, Corradi F. Diagnostic value of chest ultrasound after cardiac surgery: a comparison with chest X-ray and auscultation. J Cardiothorac Vasc Anesth. 2014 Dec;28(6):1527-32. doi: 10.1053/j.jvca.2014.04.012. Epub 2014 Sep 26. PMID 25263771
- [Background] Blaivas M, Lyon M, Duggal S. A prospective comparison of supine chest radiography and bedside ultrasound for the diagnosis of traumatic pneumothorax. Acad Emerg Med. 2005 Sep;12(9):844-9. doi: 10.1197/j.aem.2005.05.005. PMID 16141018
- [Background] Zanobetti M, Poggioni C, Pini R. Can chest ultrasonography replace standard chest radiography for evaluation of acute dyspnea in the ED? Chest. 2011 May;139(5):1140-1147. doi: 10.1378/chest.10-0435. Epub 2010 Oct 14. PMID 20947649
- [Background] Goudie E, Bah I, Khereba M, Ferraro P, Duranceau A, Martin J, Thiffault V, Liberman M. Prospective trial evaluating sonography after thoracic surgery in postoperative care and decision making. Eur J Cardiothorac Surg. 2012 May;41(5):1025-30. doi: 10.1093/ejcts/ezr183. Epub 2011 Dec 23. PMID 22219462
- [Background] Lichtenstein D, Goldstein I, Mourgeon E, Cluzel P, Grenier P, Rouby JJ. Comparative diagnostic performances of auscultation, chest radiography, and lung ultrasonography in acute respiratory distress syndrome. Anesthesiology. 2004 Jan;100(1):9-15. doi: 10.1097/00000542-200401000-00006. PMID 14695718